CLINICAL TRIAL: NCT04626089
Title: Adaptive Study for Efficacy and Safety of Metformin Glycinate for the Treatment of Patients With MS and DM2, Hospitalized With Severe Acute Respiratory Syndrome Secondary to SARS-CoV-2. Randomized, Double-Blind, Phase IIIb.
Brief Title: Metformin Glycinate in Patients With MS or DM2 , Hospitalized With COVID-19 and SARS Secondary to SARS-CoV-2
Acronym: DMMETCOV19
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Administrative decision of the company
Sponsor: Laboratorios Silanes S.A. de C.V. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: SIL-30000-II(1)
Record Dates: First submitted 2020-10-23; First posted 2020-11-12 (Actual); Last update posted 2021-04-08 (Actual); Status verified 2020-11

CONDITIONS: Severe Acute Respiratory Syndrome Coronavirus 2; Metabolic Syndrome; Type 2 Diabetes
Keywords: SARS-CoV 2; Metabolic Syndrome; Type 2 diabetes; Severe Acute Respiratory Syndrome; Metformin glycinate
MeSH Terms: conditions — Metabolic Syndrome; Diabetes Mellitus, Type 2; Severe Acute Respiratory Syndrome

STUDY DESIGN:
Intervention Model Description: Experimental group: Metformin glycinate 620 mg bid (PO) plus standard treatment for 14 days. Control Group: Placebo bid (PO) plus standard treatment for 14 days plus
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Parallel assignment experimental and placebo tablets will have same physical appearance and medicine box will be identified by kit number
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Metformin glycinate (Experimental): 620 mg bid (PO) plus standard treatment for 14 days
  Interventions: Drug: metformin glycinate
- Placebo (Placebo Comparator): Placebo tablets bid (PO) plus standard treatment for 14 days
  Interventions: Drug: Placebo oral tablet

INTERVENTIONS:
Drug: metformin glycinate — Participants randomized to metformin glycinate wil take 620 mg bid (PO) plus standard treatment for 14 days
  Other Names: DMMET
  Arms: Metformin glycinate
Drug: Placebo oral tablet — Participants randomized to placebo will take a tablet bid (PO) plus standard treatment for 14 days
  Other Names: Placebo
  Arms: Placebo

SUMMARY:
The purpose of this study is to evaluate the efficacy and safety of metformin glycinate at dose of 620 mg twice per day plus standard treatment comparing to standard treatment alone (we will use placebo) of patients who have metabolic syndrome or type 2 diabetes, which have severe acute respiratory syndrome secondary to SARS-CoV-2.

DETAILED DESCRIPTION:
After being informed about the study and potential risks, all patients will give written informed consent and undergo a 1 day screening period to determine the eligibility for study entry. At day 0, patients who meet the eligibility requirements will be randomized in a double blind (participant and investigator) in a 1:1 ratio to metformin glycinate (620 mg, taken orally twice daily) plus standard treatment or placebo (taken orally,twice daily) plus standard treatment, both will be for 14 days.

ELIGIBILITY:
Inclusion Criteria:

1. ≥ 18 years old
2. Ability to understand and the willingness to sign a written informed consent document before any study procedure
3. Metabolic syndrome or type 2 diabetes
4. Coronavirus infection, severe acute respiratory syndrome SARS-CoV- 2 confirmed by the Polymerase Chain Reaction test (PCR) ≤ 4 days before of the randomization.
5. Hospitalized patient.
6. Radiographic evidence of pulmonary infiltrates

Exclusion Criteria:

1. Participation in any other clinical trial of an experimental treatment for COVID-19
2. Evidence of multi-organ failure
3. Require mechanical ventilation before randomization
4. Pregnant patients

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2021-02 (Estimated); Primary Completion 2021-02 (Estimated); Study Completion 2021-02 (Estimated)

PRIMARY OUTCOMES:
Viral Load | Day 0 to Day 8 or patient discharge day
  Assess differences in SARS-CoV-2 viral load between participants that receive placebo vs metformin glycinate

SECONDARY OUTCOMES:
Days of supplementary oxygen if apply | Day 0 to day 28 or patient discharge day
  Assess length of supplementary oxygen
Days of supplementary mechanical ventilation if apply | Day 0 to day 28 or patient discharge day
  Assess length of mechanical ventilation
Days of Hospitalization | Day 0 to day 28 or patients discharge day
  Assess length of hospitalization
Normalization of fever | Day 0 to day 28 or patient discharge day
  Assess the difference in the Proportion of participants with normalization of fever between participants that receive placebo vs the patients with metformin glycinate
Normalization of oxigen saturation | Day 0 to day 28 or patient discharge day
  Assess the difference in the Proportion of participants with normalization of oxygen saturation between participants that receive placebo vs the patients with metformin glycinate
Number of deaths | Day 0 to day 28 or patient discharge day
  Assess the difference in the number of deaths between participants who received placebo versus the patients with metformin glycinate
Change in Serum creatinine levels | Day 0 to day 28 or patients discharge day
  Evaluate if the level increase or decrease in serum creatinine compared to baseline. units: mg/dl
Change in serum Troponin I | Day 0 to day 28 or patients discharge day
  Evaluate if the level increase or decrease in serum Creatine kinase-MB compared to baseline. Units: UI/l
Change in serum aspartate aminotransferase levels | Day 0 to day 28 or patients discharge day
  Evaluate if the level increase or decrease in serum aspartate aminotransferase compared to baseline. units: IU/l
Change in serum Creatine kinase-MB levels | Day 0 to day 28 or patients discharge day
  Evaluate if the level increase or decrease in serum Creatine kinase-MB compared to baseline. Units: UI/l
Incidence of adverse event | Day 0 to day 28 or patients discharge day
  Assess by incidence of grade 3, grade 4 and Serious adverse events

CONTACTS AND LOCATIONS:
Overall Officials: Fausto González-Villagrán, MD, Principal Investigator — Hospital Juárez de México, OPD
Locations (1):
- Hospital Juárez de México, OPD, Mexico City, Mexico

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Revert F, Ventura I, Martinez-Martinez P, Granero-Molto F, Revert-Ros F, Macias J, Saus J. Goodpasture antigen-binding protein is a soluble exportable protein that interacts with type IV collagen. Identification of novel membrane-bound isoforms. J Biol Chem. 2008 Oct 31;283(44):30246-55. doi: 10.1074/jbc.M805026200. Epub 2008 Sep 4. PMID 18772132
- [Background] Glucophage Product Monograph (metformin hydrochloride) Sanofi-Aventis Canada. Rev.28th October 2008
- [Background] NDA 20-357, Glucophage. US Food and Drug Administration. Center for Drug Evaluation and Research. Freedom of Information Office. New Drug Approval Packages. Pharmacology/Toxicology Review.
- [Background] NDA 21-842, Actoplus met. US Food and Drug Administration. Center for Drug Evaluation and Research. Freedom of Information Office. New Drug Approval Packages. Pharmacology/Toxicology Review.
- [Result] Saus J, Wieslander J, Langeveld JP, Quinones S, Hudson BG. Identification of the Goodpasture antigen as the alpha 3(IV) chain of collagen IV. J Biol Chem. 1988 Sep 15;263(26):13374-80. PMID 3417661
- [Result] Hudson BG, Tryggvason K, Sundaramoorthy M, Neilson EG. Alport's syndrome, Goodpasture's syndrome, and type IV collagen. N Engl J Med. 2003 Jun 19;348(25):2543-56. doi: 10.1056/NEJMra022296. No abstract available. PMID 12815141
- [Result] Quinones S, Bernal D, Garcia-Sogo M, Elena SF, Saus J. Exon/intron structure of the human alpha 3(IV) gene encompassing the Goodpasture antigen (alpha 3(IV)NC1). Identification of a potentially antigenic region at the triple helix/NC1 domain junction. J Biol Chem. 1992 Oct 5;267(28):19780-4. PMID 1400291
- [Result] Revert F, Penades JR, Plana M, Bernal D, Johansson C, Itarte E, Cervera J, Wieslander J, Quinones S, Saus J. Phosphorylation of the Goodpasture antigen by type A protein kinases. J Biol Chem. 1995 Jun 2;270(22):13254-61. doi: 10.1074/jbc.270.22.13254. PMID 7768924
- [Result] Borza CM, Borza DB, Pedchenko V, Saleem MA, Mathieson PW, Sado Y, Hudson HM, Pozzi A, Saus J, Abrahamson DR, Zent R, Hudson BG. Human podocytes adhere to the KRGDS motif of the alpha3alpha4alpha5 collagen IV network. J Am Soc Nephrol. 2008 Apr;19(4):677-84. doi: 10.1681/ASN.2007070793. Epub 2008 Jan 30. PMID 18235087
- [Result] Raya A, Revert-Ros F, Martinez-Martinez P, Navarro S, Rosello E, Vieites B, Granero F, Forteza J, Saus J. Goodpasture antigen-binding protein, the kinase that phosphorylates the goodpasture antigen, is an alternatively spliced variant implicated in autoimmune pathogenesis. J Biol Chem. 2000 Dec 22;275(51):40392-9. doi: 10.1074/jbc.M002769200. PMID 11007769
- [Result] Hanada K, Kumagai K, Yasuda S, Miura Y, Kawano M, Fukasawa M, Nishijima M. Molecular machinery for non-vesicular trafficking of ceramide. Nature. 2003 Dec 18;426(6968):803-9. doi: 10.1038/nature02188. PMID 14685229
- [Result] Revert F, Merino R, Monteagudo C, Macias J, Peydro A, Alcacer J, Muniesa P, Marquina R, Blanco M, Iglesias M, Revert-Ros F, Merino J, Saus J. Increased Goodpasture antigen-binding protein expression induces type IV collagen disorganization and deposit of immunoglobulin A in glomerular basement membrane. Am J Pathol. 2007 Nov;171(5):1419-30. doi: 10.2353/ajpath.2007.070205. Epub 2007 Oct 4. PMID 17916599
- [Result] Revert-Ros F, Lopez-Pascual E, Granero-Molto F, Macias J, Breyer R, Zent R, Hudson BG, Saadeddin A, Revert F, Blasco R, Navarro C, Burks D, Saus J. Goodpasture antigen-binding protein (GPBP) directs myofibril formation: identification of intracellular downstream effector 130-kDa GPBP-interacting protein (GIP130). J Biol Chem. 2011 Oct 7;286(40):35030-43. doi: 10.1074/jbc.M111.249458. Epub 2011 Aug 9. PMID 21832087
- [Result] Darris C, Revert F, Revert-Ros F, Gozalbo-Rovira R, Feigley A, Fidler A, Lopez-Pascual E, Saus J, Hudson BG. Unicellular ancestry and mechanisms of diversification of Goodpasture antigen-binding protein. J Biol Chem. 2019 Jan 18;294(3):759-769. doi: 10.1074/jbc.RA118.006225. Epub 2018 Oct 30. PMID 30377252
- [Result] Revert F, Revert-Ros F, Blasco R, Artigot A, Lopez-Pascual E, Gozalbo-Rovira R, Ventura I, Gutierrez-Carbonell E, Roda N, Ruiz-Sanchis D, Forteza J, Alcacer J, Perez-Sastre A, Diaz A, Perez-Paya E, Sanz-Cervera JF, Saus J. Selective targeting of collagen IV in the cancer cell microenvironment reduces tumor burden. Oncotarget. 2018 Jan 19;9(13):11020-11045. doi: 10.18632/oncotarget.24280. eCollection 2018 Feb 16. PMID 29541394
- [Result] Swanton C, Marani M, Pardo O, Warne PH, Kelly G, Sahai E, Elustondo F, Chang J, Temple J, Ahmed AA, Brenton JD, Downward J, Nicke B. Regulators of mitotic arrest and ceramide metabolism are determinants of sensitivity to paclitaxel and other chemotherapeutic drugs. Cancer Cell. 2007 Jun;11(6):498-512. doi: 10.1016/j.ccr.2007.04.011. PMID 17560332
- [Result] Szegezdi E, Logue SE, Gorman AM, Samali A. Mediators of endoplasmic reticulum stress-induced apoptosis. EMBO Rep. 2006 Sep;7(9):880-5. doi: 10.1038/sj.embor.7400779. PMID 16953201
- [Result] Fung TS, Liu DX. Human Coronavirus: Host-Pathogen Interaction. Annu Rev Microbiol. 2019 Sep 8;73:529-557. doi: 10.1146/annurev-micro-020518-115759. Epub 2019 Jun 21. PMID 31226023
- [Result] Catanzaro N, Meng XJ. Induction of the unfolded protein response (UPR) suppresses porcine reproductive and respiratory syndrome virus (PRRSV) replication. Virus Res. 2020 Jan 15;276:197820. doi: 10.1016/j.virusres.2019.197820. Epub 2019 Nov 16. PMID 31743697
- [Result] Schimmack G, Defronzo RA, Musi N. AMP-activated protein kinase: Role in metabolism and therapeutic implications. Diabetes Obes Metab. 2006 Nov;8(6):591-602. doi: 10.1111/j.1463-1326.2005.00561.x. PMID 17026483
- [Result] Sriwijitkamol A, Musi N. Advances in the development of AMPK-activating compounds. Expert Opin Drug Discov. 2008 Oct;3(10):1167-76. doi: 10.1517/17460441.3.10.1167. PMID 23489075
- [Result] Musi N, Hirshman MF, Nygren J, Svanfeldt M, Bavenholm P, Rooyackers O, Zhou G, Williamson JM, Ljunqvist O, Efendic S, Moller DE, Thorell A, Goodyear LJ. Metformin increases AMP-activated protein kinase activity in skeletal muscle of subjects with type 2 diabetes. Diabetes. 2002 Jul;51(7):2074-81. doi: 10.2337/diabetes.51.7.2074. PMID 12086935
- [Result] Shaw RJ, Lamia KA, Vasquez D, Koo SH, Bardeesy N, Depinho RA, Montminy M, Cantley LC. The kinase LKB1 mediates glucose homeostasis in liver and therapeutic effects of metformin. Science. 2005 Dec 9;310(5754):1642-6. doi: 10.1126/science.1120781. Epub 2005 Nov 24. PMID 16308421
- [Result] Detaille D, Guigas B, Leverve X, Wiernsperger N, Devos P. Obligatory role of membrane events in the regulatory effect of metformin on the respiratory chain function. Biochem Pharmacol. 2002 Apr 1;63(7):1259-72. doi: 10.1016/s0006-2952(02)00858-4. PMID 11960602
- [Result] Stumvoll M, Nurjhan N, Perriello G, Dailey G, Gerich JE. Metabolic effects of metformin in non-insulin-dependent diabetes mellitus. N Engl J Med. 1995 Aug 31;333(9):550-4. doi: 10.1056/NEJM199508313330903. PMID 7623903
- [Result] Otto M, Breinholt J, Westergaard N. Metformin inhibits glycogen synthesis and gluconeogenesis in cultured rat hepatocytes. Diabetes Obes Metab. 2003 May;5(3):189-94. doi: 10.1046/j.1463-1326.2003.00263.x. PMID 12681026
- [Result] Fery F, Plat L, Balasse EO. Effects of metformin on the pathways of glucose utilization after oral glucose in non-insulin-dependent diabetes mellitus patients. Metabolism. 1997 Feb;46(2):227-33. doi: 10.1016/s0026-0495(97)90307-3. PMID 9030834
- [Result] Hother-Nielsen O, Schmitz O, Andersen PH, Beck-Nielsen H, Pedersen O. Metformin improves peripheral but not hepatic insulin action in obese patients with type II diabetes. Acta Endocrinol (Copenh). 1989 Mar;120(3):257-65. doi: 10.1530/acta.0.1200257. PMID 2648723
- [Result] Tamura Y, Watada H, Sato F, Kumashiro N, Sakurai Y, Hirose T, Tanaka Y, Kawamori R. Effects of metformin on peripheral insulin sensitivity and intracellular lipid contents in muscle and liver of overweight Japanese subjects. Diabetes Obes Metab. 2008 Sep;10(9):733-8. doi: 10.1111/j.1463-1326.2007.00801.x. Epub 2007 Oct 15. PMID 17941868
- [Result] Fischer M, Timper K, Radimerski T, Dembinski K, Frey DM, Zulewski H, Keller U, Muller B, Christ-Crain M, Grisouard J. Metformin induces glucose uptake in human preadipocyte-derived adipocytes from various fat depots. Diabetes Obes Metab. 2010 Apr;12(4):356-9. doi: 10.1111/j.1463-1326.2009.01169.x. PMID 20380657
- [Result] Cataldo NA, Abbasi F, McLaughlin TL, Basina M, Fechner PY, Giudice LC, Reaven GM. Metabolic and ovarian effects of rosiglitazone treatment for 12 weeks in insulin-resistant women with polycystic ovary syndrome. Hum Reprod. 2006 Jan;21(1):109-20. doi: 10.1093/humrep/dei289. Epub 2005 Sep 9. PMID 16155076
- [Result] Cuthbertson J, Patterson S, O'Harte FP, Bell PM. Investigation of the effect of oral metformin on dipeptidylpeptidase-4 (DPP-4) activity in Type 2 diabetes. Diabet Med. 2009 Jun;26(6):649-54. doi: 10.1111/j.1464-5491.2009.02748.x. PMID 19538242
- [Result] Standeven KF, Ariens RA, Whitaker P, Ashcroft AE, Weisel JW, Grant PJ. The effect of dimethylbiguanide on thrombin activity, FXIII activation, fibrin polymerization, and fibrin clot formation. Diabetes. 2002 Jan;51(1):189-97. doi: 10.2337/diabetes.51.1.189. PMID 11756340
- [Result] Nichols GA, Gomez-Caminero A. Weight changes following the initiation of new anti-hyperglycaemic therapies. Diabetes Obes Metab. 2007 Jan;9(1):96-102. doi: 10.1111/j.1463-1326.2006.00580.x. PMID 17199724
- [Result] Landman GW, Kleefstra N, van Hateren KJ, Groenier KH, Gans RO, Bilo HJ. Metformin associated with lower cancer mortality in type 2 diabetes: ZODIAC-16. Diabetes Care. 2010 Feb;33(2):322-6. doi: 10.2337/dc09-1380. Epub 2009 Nov 16. PMID 19918015
- [Result] Gonzalez-Ortiz M, Martinez-Abundis E, Robles-Cervantes JA, Ramos-Zavala MG, Barrera-Duran C, Gonzalez-Canudas J. Effect of metformin glycinate on glycated hemoglobin A1C concentration and insulin sensitivity in drug-naive adult patients with type 2 diabetes mellitus. Diabetes Technol Ther. 2012 Dec;14(12):1140-4. doi: 10.1089/dia.2012.0097. Epub 2012 Sep 13. PMID 22974412
- [Result] JORGE GONZÁLEZ-CANUDAS, COMET GROUP Diabetes Efficacy and Safety of Metformin Glycinate vs. Metformin Hydrochloride in Metabolic Control and Inflammatory Mediators in Type 2 Diabetes Mellitus Patients. Diabetes 2019 Jun; 68(Supplement 1):
- [Result] Garza-Ocañas L, Tamez-de la O E, Iglesias-Chiesa J, Gonzalez Canudas J, Rivas-Ruiz R: Pharmacokinetics and gastrointestinal tolerability of DMMET 01 (glycinate of metformin): results of a prospective randomized trial in healthy volunteers [abstract]. Diabetes 2009;58(Suppl 1):A533.
- [Result] Granero F, Revert F, Revert-Ros F, Lainez S, Martinez-Martinez P, Saus J. A human-specific TNF-responsive promoter for Goodpasture antigen-binding protein. FEBS J. 2005 Oct;272(20):5291-305. doi: 10.1111/j.1742-4658.2005.04925.x. PMID 16218959
- [Result] Foretz M, Hebrard S, Leclerc J, Zarrinpashneh E, Soty M, Mithieux G, Sakamoto K, Andreelli F, Viollet B. Metformin inhibits hepatic gluconeogenesis in mice independently of the LKB1/AMPK pathway via a decrease in hepatic energy state. J Clin Invest. 2010 Jul;120(7):2355-69. doi: 10.1172/JCI40671. Epub 2010 Jun 23. PMID 20577053
- [Result] Rada P, Mosquera A, Muntane J, Ferrandiz F, Rodriguez-Manas L, de Pablo F, Gonzalez-Canudas J, Valverde AM. Differential effects of metformin glycinate and hydrochloride in glucose production, AMPK phosphorylation and insulin sensitivity in hepatocytes from non-diabetic and diabetic mice. Food Chem Toxicol. 2019 Jan;123:470-480. doi: 10.1016/j.fct.2018.11.019. Epub 2018 Nov 9. PMID 30414960
- [Result] Choi YH, Lee MG. Effects of enzyme inducers and inhibitors on the pharmacokinetics of metformin in rats: involvement of CYP2C11, 2D1 and 3A1/2 for the metabolism of metformin. Br J Pharmacol. 2006 Oct;149(4):424-30. doi: 10.1038/sj.bjp.0706875. Epub 2006 Aug 29. PMID 16940989
- [Result] Dianben® 1000 mg polvo para solución oral. Ficha técnica del producto. Nº de autorización de comercialización: 70545. Merck Santé S.A.S. 37 rue Saint Romain. 69008 Lyon. Francia. Fecha de revision 2010. Consultada en la web de la Agencia Española del Medicamento y de Productos Sanitarios (www.aemps.gob.es) el 27 de Marzo del 2013
- [Result] Giugliano D, De Rosa N, Di Maro G, Marfella R, Acampora R, Buoninconti R, D'Onofrio F. Metformin improves glucose, lipid metabolism, and reduces blood pressure in hypertensive, obese women. Diabetes Care. 1993 Oct;16(10):1387-90. doi: 10.2337/diacare.16.10.1387. PMID 8269798
- [Result] Landin K, Tengborn L, Smith U. Treating insulin resistance in hypertension with metformin reduces both blood pressure and metabolic risk factors. J Intern Med. 1991 Feb;229(2):181-7. doi: 10.1111/j.1365-2796.1991.tb00328.x. PMID 1900072
- [Result] Quaile MP, Melich DH, Jordan HL, Nold JB, Chism JP, Polli JW, Smith GA, Rhodes MC. Toxicity and toxicokinetics of metformin in rats. Toxicol Appl Pharmacol. 2010 Mar 15;243(3):340-7. doi: 10.1016/j.taap.2009.11.026. Epub 2010 Jan 13. PMID 20004680
- [Result] Santure M, Pitre M, Gaudreault N, Marette A, Nadeau A, Bachelard H. Effect of metformin on the vascular and glucose metabolic actions of insulin in hypertensive rats. Am J Physiol Gastrointest Liver Physiol. 2000 May;278(5):G682-92. doi: 10.1152/ajpgi.2000.278.5.G682. PMID 10801260
- [Result] Verma S, Bhanot S, McNeill JH. Antihypertensive effects of metformin in fructose-fed hyperinsulinemic, hypertensive rats. J Pharmacol Exp Ther. 1994 Dec;271(3):1334-7. PMID 7996443